CLINICAL TRIAL: NCT00412763
Title: Efficacy of Silymarin for Treatment of Acute Hepatitis In Egypt: A Randomized, Double-Blinded, Controlled Trial
Brief Title: Efficacy of Silymarin for Acute Hepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Samer S. El-Kamary, Adjunct Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-21829
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis
Keywords: Acute hepatitis; Acute viral hepatitis; Acute nonviral hepatitis; Silymarin; Milk Thistle
MeSH Terms: conditions — Hepatitis | interventions — Silymarin; milk-thistle extract

INTERVENTIONS:
Drug: Silymarin (Silybum marianum)

SUMMARY:
The overall objective of this project is to assess whether Silymarin therapy shortens illness or prevents complications in patients with acute hepatitis. We will specifically compare responses in acute hepatitis patients treated with Silymarin to those given a control preparation of a vitamin supplements in a double blinded, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
The study is designed as a double-blinded placebo controlled trial. We compare a 4 week course of therapy with silymarin tablets and a low-dose vitamin preparation (placebo) and then follow-up for a total of 8 weeks to assess treatment response. Outcomes of our randomized controlled trial are improvement in symptoms and signs, normalization of liver functions, time to resuming normal activities, and and sense of well-being. This protocol follows the standard therapeutic care for acute hepatitis except that the patients will receive either a herbal supplement (silymarin), which many patients are taking anyway, or a vitamin placebo.

Freshly collected serum will be tested for anti-HAV IgM, anti-HBc Igm, anti-HBs, HBs Ag, anti-HCV antibody, HCV-RNA, anti-HDV IgM, anti-HEV IgM, CMV and EBV and for alanine aminotransferase (ALT), AST, direct and total bilirubin.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the fever hospital and presenting with symptoms and signs that may be consistent with a diagnosis of acute hepatitis.
* Recent (<1 month) history of illness.
* Elevation of ALT > 2.5 normal.
* At least 13 years old.

Exclusion Criteria:

* History suggestive of severe drug-induced acute hepatitis.
* Children 12 years and younger.
* Pregnant or breastfeeding women
* Suspected hypersensitivity to Silymarin or vitamin preparations.
* Evidence of advanced liver disease e.g. history or presence of ascitis, bleeding esophageal varices, and hepatic encephalopathy.
* Patients who are critically ill, with multisystem failure or cancer.
* Substance abuse such as IV drugs.
* Any other conditions, which in the opinion of the investigator would make the patient unsuitable for enrollment or could interfere with the patient's participation in and completion of the protocol.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2003-07; Study Completion 2005-10

PRIMARY OUTCOMES:
Primary outcomes were symptoms and signs of acute hepatitis and results of liver function tests on days 3, 5 and 7 in the hospital and in the outpatient clinic at weeks 2, 4, and 8.

SECONDARY OUTCOMES:
Side-effects and adverse events were ascertained by self-report on days 3, 5 and 7 in the hospital and in the outpatient clinic at weeks 2, 4, and 8. .

CONTACTS AND LOCATIONS:
Overall Officials: George T Strickland, MD, PhD, Principal Investigator — University of Maryland, Baltimore